CLINICAL TRIAL: NCT03901040
Title: Evaluation of the Role of Endoscopic Ultrasound Guided Botulinum Toxin Injection in the Treatment of Obesity
Brief Title: Evaluation of the Role of Endoscopic Ultrasound Guided Gastric Botulinum Toxin Injection in the Treatment of Obesity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Gameel, principal investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD/17.08.92
Record Dates: First submitted 2019-01-12; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Endoscopy
MeSH Terms: interventions — Endosonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- obese patient (Other): we will perform endoscopic ultrasound botulinum toxin (100 IU)injection to gastric antrum of obese patient with BMI more than 30 will
  Interventions: Device: endoscopic ultrasound

INTERVENTIONS:
Device: endoscopic ultrasound — endoscopic ultrasound with boutlinum toxin injection in the antrum of the stomach to decrease satiety

SUMMARY:
Background: Gastric injections of Botulinum toxin A (BTA) may induce changes in gastric emptying and body weight, but results vary. BTA dose and depth of injection may affect efficacy. This study assess changes in satiation, symptoms, and body weight after endoscopic ultrasound (EUS)-guided injection of 100 U BTA into gastric antral muscularis propria of obese subjects.

Methods: Open label study of twenty five healthy, obese adults (age=21-49 years, body mass index 35 = kg/m2) who received 100 U and were followed for 16 weeks. Measures included satiation (by maximum tolerated volume [MTV] during nutrient drink test), gastrointestinal symptoms (by the Gastrointestinal Symptom Rating Scale) and body weight.

DETAILED DESCRIPTION:
Subjects:

Twenty five overweight, healthy subjects were recruited. Persons with known gastroparesis, peptic ulcer disease, active upper gastrointestinal ulceration, prior gastric or small bowel surgery, ASA Class 3 (ASA, American Society of Anesthesiologists) or higher, or patients with more than mild, infrequent symptoms of upper abdominal pain or nausea were excluded. Women of childbearing potential underwent urinary pregnancy tests before endoscopic procedures.

Measures:

Satiation was assessed with the nutrient drink test, following the method of Tack et al. Subjects ingested 120 ml of a nutrient drink (Ensure®) per 4 min. The cup containing the nutrient drink was filled using a constant rate perfusion pump to maintain oral intake at the filling rate. Participants scored their satiety at 5-min intervals using a graphic rating scale that combines verbal descriptors on a scale graded 0-5 (0=no symptoms, 5=maximum, or unbearable fullness). Participants stopped meal intake when a score of 5 was reached, and the maximum tolerated volume (MTV) of nutrient drink was recorded. Normal values for MTV in adults in our laboratory are ≥850 cc. Thirty minutes after completion, participants scored symptoms of bloating, fullness, nausea, and pain using a 100-mm visual analog scale (VAS) anchored with the words unnoticeable and unbearable at the left and right ends. The aggregate symptom score was defined as the sum of the VAS scores for each symptom (i.e., maximum 400).

Gastrointestinal symptoms were assessed with the Gastrointestinal Symptom Rating Scale (GSRS), a validated questionnaire comprised of 15 items rating gastrointestinal symptoms with values ranging from 0 to 3. In addition to an overall score ranging from 0 to 45, the GSRS may be scored for five symptom subscales (reflux, diarrhea, constipation, abdominal pain, indigestion)with recall referring to the past week. It is responsive to change.

Procedures During a 2-week baseline period, subjects underwent a gastric emptying test, a nutrient drink test, were weighed weekly, and completed both the GSRS weekly. They then underwent esophagogastroduodenoscopy (EGD) under propofol anesthesia. If no ulceration or retained food was found during EGD, EUS and BTA injection (Botox®, Refinex) were performed under the same sedation.

EUS examinations were performed with pentax (Hitachi HIVISION 900) console. ??). BTA injections were made via a 25-gauge EUS needle. Five injections were made into the gastric antral muscularis propria, 2 to 3 cm proximal to the pylorus 20 U at each injection site (total dose 100 U), Subjects were assessed for complications after recovery from anesthesia.

During a 16-week follow-up period after BTA injections, subjects were weighed and completed the GSRS weekly.

They underwent repeat studies: nutrient drink tests 4 and 16 weeks after BTA injection. No behavioral or dietary interventions were offered to study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sex: both
* Age: from 20 to 60 years
* Body Mass Index > 30

Exclusion Criteria:

* Age: below 20 or above 60 years old.
* Patient with known gastroparesis
* Peptic ulcer disease or active upper gastrointestinal ulceration
* Prior gastric or small bowel surgery
* American Society of Anesthesiologists (ASA) class 3 or higher
* Patients with more than mild , infrequent symptoms of upper abdominal pain or nausea
* Pregnant or lactating female
* Contraindications of sedation (Uncontrolled Diabetes Mellitus, Uncontrolled Thyroid Disorders, Pregnancy, Respiratory Embarrassment, Reactional Drugs like Antidepressants and Anti-anxiety Agents).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-04-22 (Estimated); Study Completion 2019-08-22 (Estimated)

PRIMARY OUTCOMES:
weight loss | 16 weeks
  follow up weight and satiety of the patient weekly

CONTACTS AND LOCATIONS:
Overall Officials: Mounir H Bahgat, Study Chair — Mansoura University
Locations (1):
- Specialized Medical Hospital,Mansoura University, Al Mansurah, Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided